CLINICAL TRIAL: NCT03651492
Title: Effects of Nocturnal Hypertension on Sleep Quality in Renal Transplant Recipients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Federico II University (Other)
Responsible Party: Principal Investigator, Massimo Sabbatini, Associate Professor of Nephrology, Federico II University
Other Study IDs: FedericoIIUniversity
Record Dates: First submitted 2018-08-17; First posted 2018-08-29 (Actual); Last update posted 2018-08-29 (Actual); Status verified 2018-08

CONDITIONS: Hypertension; Nephropathy; Renal Transplant; Sleep Disorder
Keywords: nocturnal hypertension; renal transplantation; sleep quality
MeSH Terms: conditions — Hypertensive Nephropathy; Sleep Wake Disorders; Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: questionnaire administration — All the patients will be administered the Pittsburgh Questionnaire after completion of ABPM.

SUMMARY:
Nocturnal hypertension (i.e. blood pressure values >120/70 or 10% higher than diurnal values, as measured by ambulatory blood pressure monitoring, ABPM) is particularly frequent in renal transplant recipients (RTR), despite the use of antihypertensive drugs. Since RTR are also affected by several sleep disorders (like insomnia, restless legs syndrome, sleep apnoea) that frankly impair their quality of sleep (SQ), the aim of the present study is to ascertain whether a relationship exists between nocturnal hypertension and SQ. In fact, both nocturnal hypertension and sleep disorders may favour the onset or the progression of cardiovascular diseases, the first cause of death in RTR.

DETAILED DESCRIPTION:
Hypertension affects the great majority of renal transplant recipients (RTR) and its persistence may negatively influence the outcome of the graft. Unfortunately, its diagnosis is not univocal since office measurement of blood pressure (BP) may reveal a "white coat hypertension" in normotensive subjects, or might not detect hypertension if pills are taken immediately before BP control. Therefore for a correct diagnosis the use of ambulatory BP monitoring (ABPM) is strongly advised. Recent studies employing this methodology have shown that the prevalence of nocturnal hypertension (i.e. blood pressure values >120/70 or 10% higher than diurnal values) affects a great number of renal transplant recipients (RTR), even despite the use of antihypertensive drugs ("non-dipper" patients). It is well known that nocturnal hypertension enhances the development of cardiovascular diseases, but it is not clear whether (and to what extent) it also affects the quality of sleep of these patients. Sleep disturbances like insomnia, restless legs syndrome and sleep apnoea, in fact, are particularly common in RTR, despite these patients report significantly better quality of life compared to patients with chronic renal failure under conservative or dialysis treatment. The working hypothesis of the present study is to evaluate whether any relationship exists between nocturnal hypertension and sleep quality, since also sleep disorders may favour the onet and the progression of cardiovascular diseases, the first cause of death in RTR with functioning graft.

The study will be carried out on all the available RTR in regular follow-up at the DH of Nephrology and Renal Transplantation of the University Federico II of Naples (Italy). Inclusion criteria are: age >18 years, renal transplant vintage >1 year, stable renal function in the last 6 month, no change in immunosuppressive nor antihypertensive treatment in the last 3 months, no intercurrent infection in the last 3 months. Twenty-four hour ABPM will be performed during the regular follow-up of patients in the investigator's Unit. Hypertension will be diagnosed when the patient takes antihypertensive drugs or when his . BP is >130/80 mmHg (24-hour average value), or >135/85 (average values of daily BP) or >120/70 (average values of nocturnal BP). The patient will be considered "non-dipper" when the ratio Systolic nocturnal BP/Systolic diurnal BP is >0.9.

Sleep quality will be evaluated through a validated version of the Pittsburgh Sleep Questionnaire a self-rated questionnaire, consisting of 19 questions which assess a wide variety of factors relating to sleep quality, including estimates of sleep duration and latency and of frequency and severity of specific sleep-related problems. These 19 items are grouped into seven-component scores, each weighted equally on a 0-3 scale. The seven components are then summed to yield a global index (PSQI) ranging between 0 and 21; higher scores indicate a worse sleep quality (>5, poor sleepers; <5, good sleepers). The seven components of the PSQI are subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbances, use of sleeping medications, and daytime dysfunction. The relationship between nocturnal hypertension and sleep quality will be evaluated either by bivariate analysis and by multiple linear regression analyses. In the multivariate model, all the variables associated to an elevated night/day systolic pressure ratio will be considered if the P value is 0.10 or less at bivariate analysis. The relationship between increased night/day SBP ratio and increased PSQI will be also investigated by multivariate logistic regression model.

ELIGIBILITY:
Inclusion Criteria:

* Age>18 years
* Transplant vintage >1 year;
* Stable renal function in the last 6 months;
* No change in antihypertensive and immunosuppressive therapy in the last 3 months;
* No rejection episode in the last 6 months.

Exclusion Criteria:

* Intercurrent infections in the last 3 months;
* Treatment with sleeping or antidepressant pills;
* Patients with neurological problems in treatment with drugs acting on central nervous system;
* Patients unable to understand the meaning of the questions.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with functioning renal transplantation in regular follow-up at DH of renal transplantation of the University Federico II of Naples (Italy)
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2017-06-01 (Actual); Primary Completion 2019-06-01 (Estimated); Study Completion 2020-01-31 (Estimated)

PRIMARY OUTCOMES:
Prevalence of "poor sleepers", as assessed by Pittsburgh Questionnaire, among renal transplant recipients with elevated blood pressure, measured by ambulatory continuous monitoring. | Given the cross-sectional nature of the study, there is a single determination of sleep quality in each patient, carried out after completion of 24-hour ABPM, during a scheduled follow-up visit.
  Sleep quality will be evaluated by the Pittsburgh Questionnaire, which allows to investigate on 7 different components of sleep, determining a score ranging between 0 and 19: a score>5 defines a "poor sleeper". Through bivariate and multivariate analysis, the study will evaluate which relationship exists between nocturnal hypertension ands sleep quality.

CONTACTS AND LOCATIONS:
Locations (1):
- University Federico II, Napoli, Italy

IPD SHARING:
Plan to Share IPD: No